CLINICAL TRIAL: NCT02937246
Title: Efficacy of Partial Covered Double Bare Metal Stent Compared to Uncovered Double Bare Metal Stent in Malignant Biliary Obstruction: A Multicenter Prospective Randomized Trial
Brief Title: Efficacy of Partial Covered Double Bare Metal Stent Compared to Uncovered Double Bare Metal Stent in Malignant Biliary Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-1147
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- the intervention group (Experimental): Partial covered double bare metal stent
  Interventions: Device: SEMS(self-expandable metallic stent)
- the control group (Active Comparator): Uncovered double bare metal stent
  Interventions: Device: Stenting by ERCP (endoscopic retrograde cholangiopancreatography)

INTERVENTIONS:
Device: SEMS(self-expandable metallic stent) — Find the obstruction site by ERCP(endoscopic retrograde cholangiopancreatography) and insertion the SEMS(self-expandable metallic stent) through duodenal endoscopy. Metal stents are inserted to ensure adequate decompression and bile drainage. The diameter and stent lengths can be changed according to the lesion.
  Other Names: Obstructive jaundice decompression with endoscopic metal stenting
  Arms: the intervention group
Device: Stenting by ERCP (endoscopic retrograde cholangiopancreatography)
  Arms: the control group

SUMMARY:
Previous studies indicated that covered stents are less likely to become occluded in comparison to bare stents. While the probability of occlusions caused by tumor in-growth is less in covered stents, they are more likely to spontaneously migrate to a position that is distal to the original deployment site. However, newer covered stents with improved designs, such as the partially covered double bare metallic stent used for this study, include features to mitigate the migration issue. The purpose of this study is to confirm whether the difference in patency rate between regular covered stents and bare stents, which has already been well established by existing studies, is also reproducible when double covered stents are compared against double bare stents.

DETAILED DESCRIPTION:
Malignant obstructive jaundice is a common complication of advanced stage cholangiocarcinoma, GB cancer, and pancreatic cancer. In biliary stricture by malignancy, biliary drainage with placement of self-expanding metal stent (SEMS) for palliation is the therapy of choice in these patients. When compared to plastic stents, SEMS present a significantly decreased risk of recurrent biliary obstruction. SEMS are also more cost-effective than plastic stents in patients with a life expectancy of longer than 4 months. However, despite their numerous benefits, SEMS become occluded in up to 50 % of patients in the first 6-8 months. In order to minimize the occurrence of this issue, covered stents were developed. Previous studies indicated that covered stents are less likely to become occluded in comparison to bare stents. While the probability of occlusions caused by tumor in-growth is less in covered stents, they are more likely to spontaneously migrate to a position that is distal to the original deployment site. However, newer covered stents with improved designs, such as the partially covered double bare metallic stent used for this study, include features to mitigate the migration issue. The purpose of this study is to confirm whether the difference in patency rate between regular covered stents and bare stents, which has already been well established by existing studies, is also reproducible when double covered stents are compared against double bare stents.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed malignant biliary obstruction or clinically defined malignant biliary obstruction
* malignant biliary obstruction was located more than 1cm from the hilum
* older than 20 years old
* Life expectancy > 6 months
* Inoperable case due to advanced stage or comorbidity
* Informed consent obtained

Exclusion Criteria:

* Inadequate case for ERCP
* Failed endoscopic approach to duodenum or biliary tract
* biliary obstruction was located at hilum or IHD
* patients with uncontrolled infection
* Pregnancy
* No signed informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Mean duration of stent patency | 6 months after stenting
  Check the duration until the date of obstruction of inserted stent within 6 months after stenting

SECONDARY OUTCOMES:
Patency rate of stent | 6 months after stenting
Overall survival | 6 months after stenting

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SW, Lee KJ, Chung MJ, Jo JH, Lee HS, Park JY, Park SW, Song SY, Kang H, Kim EJ, Kim YS, Cho JH, Bang S. Covered versus uncovered double bare self-expandable metal stent for palliation of unresectable extrahepatic malignant biliary obstruction: a randomized controlled multicenter trial. Gastrointest Endosc. 2023 Jan;97(1):132-142.e2. doi: 10.1016/j.gie.2022.08.041. Epub 2022 Sep 7. PMID 36084714